CLINICAL TRIAL: NCT06652815
Title: Cognition, Metacognition, and Stigma in Patients With Suicidal Ideation
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Other Study IDs: STUDY23010161; D43TW009114 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Persons With High Suicide Ideation or Attempts
Keywords: Suicide attempt; Metacognition; suicide ideation; Executive function
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with suicide attempt or suicide ideation: Individuals with high suicide ideation or suicide attempts visiting ABVIMS -Dr. RML Hospital for treatment will be screened for this study.
  Interventions: Behavioral: Suicide ideation or suicide attempt

INTERVENTIONS:
Behavioral: Suicide ideation or suicide attempt — Individuals with high suicide ideation or suicide attempts visiting ABVIMS -Dr. RML Hospital for treatment will be screened for this study. socio- demographics details will also be gathered. Following this Depression, Anxiety and Stress Scale (DASS-21), Wisconsin Card Sorting Test (WCST), Metacognitions Scale (MCQ-30) and Stigma of Suicide Scale (SOSS) will be administered.

SUMMARY:
Deficits of executive function, meta cognition and stigma is known in suicidal ideation; however, their relationship is unknown. Since many studies use a single indicator of executive function and, it was considered important to study. Metacognition, executive functioning and stigma are the possible driving force behind the suicidal behavior in human being. With respect to research in the Indian context, there is paucity of studies exploring these factors. The purpose of the present study is to explore the relationships between executive functioning, metacognition, and stigma in suicidal ideation and suicide attempters in the Indian setup, where there is a lacuna in research regarding the same. Having a detailed understanding of these psychological parameters will be helpful in suicide prevention and management.

DETAILED DESCRIPTION:
Worldwide 10 to 20 million individuals attempt suicide every year. The suicide rate in India is 10.3. In the last three decades, the suicide rate has increased by 43% but the male female ratio has been stable at 1.4: 1. Majority (71%) of suicide in India are by persons below the age of 44 years which imposes a huge social, emotional and economic burden. Those having suicide ideas, about one third of them act with a suicide attempt, and 60% of these transitions occur within the first year after onset of suicidal thoughts.

Executive functioning and Suicide Studies reported that deficits in some executive functions are correlated with an elevated risk for suicide attempts. Executive dysfunction may interfere with an individual's ability to understand that they are at risk for suicide as well as with their ability to cope with that risk. Although past studies have identified the role of cognitive factors in suicide, little has been done to explore the cognitive processes involved in suicidal thinking in adults (Ong et al. 2016). Neuropsychological alterations can lead to inaccurate perception, interpretation, and response to environmental information, which could be a risk factor for suicide (Fernández-Sevillano et al. 2021).

Metacognition is an essential process regarding decision making and coping with stressful life events. It describes the awareness of person's cognitions in relation to suicide (thoughts, beliefs and attributions). The suicidal person feels helpless and decides that death is only solution. The person has narrowed all his/her options solely to death. Knowing these patterns will give some guidance in talking to a suicidal person. It is significant for assessing to try to accept and understand feelings "meta-emotion" and thought/attributions "meta-cognition" the person is expressing (Abdulla et al. 2018).

Stigma is most often defined as a mark of disgrace or infamy; a stain or reproach, as on one's reputation. In suicide investigators talk about public and self-stigma. Both forms of stigma can separately cause social isolation, demoralization, hopelessness and other consequences that interfere with the previous functioning. Because of the high incidence of psychological changes after stigma it is crucial for the bereaved to have close mental health services. But stigma is a barrier to treatment seeking. After suicide attempt most survivors feel stigmatized but it is not yet known which factors modify the perception of stigma (Sabina et al. 2017).

The purpose of the present study is to explore the relationships between executive functioning metacognition, and stigma in suicidal ideation and suicide attempters in the Indian setup, where there is a lacuna in research regarding the same.

Research questions

* What is the executive functioning, metacognitive beliefs, and stigma in persons with high suicide ideation or attempts?
* Is there any relationship among executive functioning, metacognitive beliefs, and stigma in these individuals? Hypotheses There will be a relationship among executive functioning, metacognitive beliefs, and stigma in persons with high suicide ideation or attempts.

Objective To assess the executive functioning, metacognitive beliefs, and stigma in persons with high suicide ideation or attempts.

To study the relationship among executive functioning, metacognitive beliefs, and stigma in persons with high suicide ideation or attempts.

Methodology Samples size: Total number of sample for this study will be N=212. The sample size 212 was calculated on the basis of estimated population of 1000 using Epitools online sample size calculator (https://epitools.ausvet.com.au/oneproportion) , and Confidence level was 0.95, with Desired precision of estimate=0.05.

Sampling: Probability sampling (Simple random sampling (Every Individual with high suicide ideation or suicide attempts visiting to ABVIMS -Dr. RML Hospital for treatment will be screened for this study.

The present study is a cross sectional study. For the purpose of this study, individuals with suicidal ideation and attempts who are seeking treatment at the outpatient department of Psychiatry, as well as medical emergency of Dr. RML Hospital or referred to Department of Clinical Psychology would be approached to participate in the study.

After establishing the rapport, diagnostic clarifications (ICD-10) and screening for high suicide ideation using Beck Scale for Suicidal Ideation (BSSI), inclusion and exclusion criteria will be applied. Participant who fulfils inclusion criteria will be introduced to the study details, then they will be explained about the purpose of the study and its associated aspects and informed consent will be taken. Their socio- demographics details will also be gathered. Following this Depression, Anxiety and Stress Scale (DASS-21), Wisconsin Card Sorting Test (WCST), Metacognitions Scale (MCQ-30) and Stigma of Suicide Scale (SOSS) will be administered.

All the data will be kept confidential in lock and key and using password protected files. Once all the assessment will be completed data entry in excel sheets will be done and analysis of the data will be done using appropriate SPSS statistical package. After all the analysis completed result and discussion of the study will be prepared.

Detail of tools to be used:

1. ICD-10 Research diagnostic criteria
2. Socio-demographic and clinical data sheet
3. Depression, Anxiety and Stress Scale-21 Items (DASS-21)
4. Beck Scale for Suicidal Ideation (BSSI)
5. Wisconsin Card Sorting Test (WCST)
6. Metacognitions Scale (MCQ-3)
7. Stigma of Suicide Scale (SOSS)

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Age between 18 to 60 years.
* Able to read and write in Hindi and English
* With a primary mental health diagnosis of anxiety, depression, acute stress reaction or adjustment disorder, or with no diagnosis at all
* Persons with high suicidal ideation (Score 2 or more in first five items of BSSI)
* Person who attempted suicide in last three months.

Exclusion Criteria:

* Any comorbid personality disorder diagnosis
* Diagnosis of a major mental disorder such as Schizophrenia or Bipolar Affective Disorder.
* Intellectual Disability and neurological disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The present study is a cross sectional study. For the purpose of this study, individuals with suicidal ideation and attempts who are seeking treatment at the outpatient department of Psychiatry, as well as medical emergency of Dr. RML Hospital or referred to Department of Clinical Psychology would be approached to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Metacognition measured by Metacognitions Questionnaire (MCQ-3) scores | Within one week
  The Metacognitions Questionnaire-30 (MCQ-30) is a self-report measure that assesses metacognitive beliefs. The MCQ-30 is comprised of five factors. Responses are required on a four-point scale ranging from 1 (do not agree) to 4 (agree very much), high scores reflect more reported problems with the item in question.
Depression, Anxiety and Stress Scale-21 scores | Within one week
  Depression, Anxiety and Stress Scale-21 Items (DASS-21): The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.Higher scores mean more anxiety or depression and low scores means low anxiety or depression.
Stigma of Suicide Scale (SOSS) scores | Within one week
  The Stigma of Suicide Scale is designed to assess stigmatizing attitudes of general community members toward people who suicide. The short form consists of 16 items. Each item consists of a one-word descriptor of a person who dies by suicide. We will use the short form. Each item is to be rated on a 5-point Likert scale from (1) strongly disagree to (5) strongly agree. Higher scores indicate higher levels of stigma towards people who suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the trial as well as protocol will be shared on request at 1-2 years after article publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After one year of publication of results of the study.
Access Criteria: Study should be ethically approved and scientifically sound.